CLINICAL TRIAL: NCT01604421
Title: Randomized Evaluation of the Use of Plastic Bags to Prevent Neonatal Hypothermia in Developing Countries-Part II
Brief Title: Evaluation of Use of Plastic Bags to Prevent Neonatal Hypothermia-Part II
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no personnel available to enroll patients- decision made to not complete study
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Children's Health System, Alabama (Other)
Responsible Party: Principal Investigator, Wally Carlo, Edwin M. Dixon Professor of Pediatrics, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UAB Neo 007
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Hypothermia
Keywords: Hypothermia; Low birth weight; Newborn; Plastic bag; Thermoregulation
MeSH Terms: conditions — Hypothermia | interventions — Body Temperature Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thermoregulation-standard care (Sham Comparator): Standard thermoregulation without a plastic bag from one hour after birth until discharge or 24 hours after birth, whichever comes first.
  Interventions: Procedure: Thermoregulation-standard care
- Thermoregulation-with plastic bag (Active Comparator): Thermoregulation with plastic bag covering torso and lower extremities from one hour after birth until discharge or 24 hours after birth to assist with thermoregulation. The infant's axillary temperature will be monitored for 24 hours or until discharge, whichever comes first.
  Interventions: Procedure: Thermoregulation with plastic bag

INTERVENTIONS:
Procedure: Thermoregulation-standard care — Standard care without plastic bag. One hour after birth, a blanket will be wrapped around the infant and he/she will receive a wool hat, according to standard practices. The infant's axillary temperature will be monitored for 24 hours or until discharge, whichever comes first.
  Arms: Thermoregulation-standard care
Procedure: Thermoregulation with plastic bag — One hour after birth, the infant will be placed into a plastic bag up to his/her axillae, and the bag will be folded and taped to itself to prevent it from covering the infant's nose or mouth. A blanket will be wrapped around the infant, and he/she will receive a wool hat. The infant will remain in the bag, which will be changed when soiled, for 24 hours or until discharge, whichever occurs first.
  Arms: Thermoregulation-with plastic bag

SUMMARY:
The overall hypothesis is that plastic bags used in combination with WHO thermoregulation care will reduce the incidence of hypothermia in preterm/low birth weight and full term infants when compared to routine WHO thermoregulation care alone. Part II is for preterm/low birth weight infant with or without plastic head cover used from 1 hour after birth until discharge or 24 hours after birth to assist with temperature regulation.

DETAILED DESCRIPTION:
Due to limited resources, hospitals in the developing world struggle to provide sufficient incubators and to maintain climate-controlled nurseries. Therefore, premature low birth weight infants continue to be at an increased risk of hypothermia throughout their hospitalizations. This study will compare the incidence of hypothermia in preterm/low birth weight infants randomized to receive WHO thermoregulation care (control groups) or WHO thermoregulation care and a plastic bag covering their torsos and lower extremities (intervention group) starting at one hour after birth and continued to discharge or 24 hours after birth, whichever occurs first. The axillary temperature of each infant will be taken one hour after birth, every subsequent 3-4 hours, and at discharge or 24 hours after birth when infants will be removed from the plastic bags. Seizures, hyperthermia, room temperature, and death will be recorded throughout the hospitalization for all infants. With an estimated baseline hypothermia rate of 50% and a hypothesized 20% absolute risk reduction (40% relative risk reduction), a sample size of 182 will be used to have a power of 80% and a confidence interval of 95%.

ELIGIBILITY:
Inclusion Criteria:

* Estimated gestational age 29-36 6/7 weeks or birth weight 1400-2500g
* Delivery in the hospital

Exclusion Criteria:

* Infant admitted to the NICU
* Birth weight less than 1400 gms
* Abdominal wall defect or myelomeningocele
* Major congenital anomalies
* Blistering skin disorder

Ages: 1 Hour to 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-02 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Axillary temperature < 36.5 degrees Celsius | Discharge or 24 hours after birth
  Temperature taken per axilla at one hour after birth. Temperatures 36.0-36.4 will be classified as mild hypothermia, 32.0-35.9 will be classified as moderate hypothermia, and <32.0 as severe hypothermia.

SECONDARY OUTCOMES:
Seizure | Up to 4 weeks
  Seizure activity diagnosed by medical director or nurse. No electroencephalogram will be done.
Respiratory Distress Syndrome (RDS) | Up to 4 weeks
  Documentation of increased work of breathing, retractions, and a need for oxygen, intubation, or surfactant
Pneumothorax | Up to 4 weeks
  Either chest radiograph documentation or clinical deterioration consistent with air leak
Sepsis | Up to 4 weeks
  Culture proven or culture negative clinically treated course consistent with sepsis
Necrotizing enterocolitis or intestinal perforation | Up to 4 weeks
  Documentation of pneumatosis or intestinal perforation on x-ray or treatment course for clinical necrotizing enterocolitis per Bell's Classification stage greater than 1.
Death | Up to 4 weeks
  Cardiorespiratory failure
Hyperthermia | Up to 4 weeks
  Axillary temperature > 38 degrees Celsius per temperature taken per axilla for one minute
Temperature and humidity | 1-72 hours after birth
  A recording of the room temperature and humidity will be obtained with each axillary temperature measurement

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University Teaching Hospital, Lusaka, Zambia